CLINICAL TRIAL: NCT06873412
Title: The Regulatory Effect of Probiotics-Polygonatum Sibiricum on Liver Health and Metabolic Disorders in Middle-Aged and Elderly People: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Effects of Compound Probiotics-Polygonatum Sibiricum on Liver Health and Metabolism in Middle-aged and Elderly People
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20250302
Record Dates: First submitted 2025-03-02; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Intervention group of polygonatum-probiotics complex, take 1 piece (2.0 g) daily
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): maltodextrin, take 1 piece (2.0 g) daily
  Interventions: Dietary Supplement: Placbo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of the study will last for 3 months, and each subject will be followed up 3 times (month 0, Month 1, Month 2, month 3).
  Arms: Probiotic group
Dietary Supplement: Placbo — The experimental phase of the study will last for 3 months, and each subject will be followed up 3 times (month 0, Month 1, Month 2, month 3).
  Arms: Placebo group

SUMMARY:
The purpose of this study was to evaluate the regulatory effects of Huangqian-biobacteria compound preparation on liver health and related metabolic disorders in middle-aged and elderly people, observe its effects on liver function indexes, basal metabolic rate, markers of oxidative stress, inflammatory factors and intestinal microecology, and evaluate the incidence of adverse reactions in subjects during the 3-month intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subjects is 40-80 years old; 2. The subject meets one of the following metabolic disease components: ① abdominal B - ultrasound shows fatty liver or fat infiltration; ② arterial blood pressure is higher than 130/85mmHg, or the subject is on antihypertensive treatment; ③ prediabetes or type 2 diabetes, with fasting blood glucose above 6.1mmol/L; ④ overweight or obesity, with BMI of 24.0kg/m² or more, or male waist circumference of 90cm or more, female waist circumference of 85cm or more, or excessive body fat content and percentage.

-

Exclusion Criteria:

1. People who are allergic to any of the pharmaceutical ingredients used in this study; A history of alcohol abuse (drinking more than 14 units of alcohol per week :1 unit = 285mL for beer, 25mL for spirits, 100mL for wine);
2. Patients who received probiotics within 1 month before taking the experimental drug;
3. Recent history of gastrointestinal bleeding, obstruction, perforation, tumor and other serious organic diseases;
4. Aminotransferase index > 3 times the normal value;
5. Kidney disease (creatinine index higher than normal);
6. Patients with serious psychological and mental diseases, resulting in the inability to express themselves normally;
7. Patients with infectious liver diseases, such as hepatitis B and C;
8. The female subject is breastfeeding or has a positive pregnancy test result during the screening period or during the test -

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in alanine aminotransferase (ALT) levels | 3 months
  ALT level decline indicates improved liver function, assessed via blood tests.
Changes in aspartate aminotransferase (AST) levels | 3 months
  AST level decline indicates improved liver function, assessed via blood tests.

SECONDARY OUTCOMES:
Changes in basal metabolic rate | 3 months
  The Mifflin-St Jeor equation was used to evaluate the subject's basal metabolic level, reflecting the body's energy expenditure at rest.
Metabolic index | 3 months
  Blood pressure: Evaluate the effects of the tested product on age-related cardiovascular health and monitor changes in systolic and diastolic blood pressure.
Gamma-glutamyltransferase (GGT) | 3 months
  Evaluate the effects of the tested product on liver-related components. GGT: The unit is U/L.
Total bilirubin (TBil) | 3 months
  Evaluate the effects of the tested product on liver-related components. TBil: Unit: μmol/L.
Uric acid | 3 months
  Evaluate the effects of the tested product on liver-related components. Uric acid: unit: μmol/L.
Weight | 3 months
  Evaluate the effects of the tested product on body weight. Weight: Unit: kg.
BMI (body mass index) | 3 months
  The effects of the product on body mass index were evaluated. BMI: Unit: kg/m².
Fasting blood glucose | 3 months
  Evaluate the effect of the tested product on blood sugar levels. Fasting blood glucose: the unit is mmol/L.
Total cholesterol | 3 months
  The effect of the tested product on lipid levels was evaluated. Total cholesterol: Unit: mmol/L.
Triglyceride | 3 months
  The effect of the tested product on lipid levels was evaluated. Triglyceride: The unit is mmol/L.
Low-density lipoprotein (LDL) | 3 months
  The effect of the tested product on lipid levels was evaluated. LDL: The unit is mmol/L.
High density lipoprotein (HDL) | 3 months
  The effect of the tested product on lipid levels was evaluated. HDL: The unit is mmol/L.
Changes in malondialdehyde (MDA) levels | 3 months
  Evaluate the effects of test products on oxidative stress levels. MDA: The unit is μmol/L.
Changes in the level of superoxide dismutase (SOD) | 3 months
  Evaluate the effects of test products on oxidative stress levels. SOD: The unit is U/mL.
Changes in glutathione (GSH) levels | 3 months
  Evaluate the effects of test products on oxidative stress levels. GSH: Unit: μmol/L
Fatigue Severity Scale (FSS) | 3 months
  Evaluate the fatigue severity of the tested product. FSS score: The unit is points, ranging from 1 to 7 points.
  1 score: No fatigue Score 7: Extreme fatigue Higher score: indicates more severe fatigue
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  Participants' overall sleep quality over the past three months was assessed. PSQI score: The unit is points, ranging from 0 to 21 points. 0 score: Best sleep quality 21 points: worst sleep quality Higher score: indicates poorer sleep quality
Short-chain fatty acids (SCFAs) | 3 months
  hort-chain fatty acids: Short-chain fatty acids such as acetic acid, propionic acid, and butyric acid are analyzed in stool samples by gas chromatography-mass spectrometry (GC-MS) or high performance liquid chromatography (HPLC).
  Acetic acid: unit: μmol/g fecal matter. Propionic acid: The unit is μmol/g feces. Butyric acid: The unit is μmol/g feces.
Fecal flora structure (16S rRNA sequencing) | 3 months
  16S rRNA sequencing: Bacterial 16S rRNA genes in fecal samples are analyzed by high-throughput sequencing techniques to determine the diversity and composition of the gut microbiota.
  Diversity index: such as Shannon index, Chao1 index, etc., used to measure the diversity of flora.
  Composition analysis: The relative abundance of major bacterial phyla, genera and species is determined by taxonomic analysis.
Inflammatory factor | 3 months
  Changes in serum levels of inflammatory cytokines (IL-6, IL-1β, TNF-α, IP-10) : To evaluate the effect of the tested product on the inflammatory response and reflect the immune status of the body.
Fatty liver morphology | 3 months
  Abdominal B-ultrasound: To evaluate the effect of the tested product on the morphology of fatty liver, reflecting the liver fat deposition.